CLINICAL TRIAL: NCT06353412
Title: Evaluation of the Current Treatment Methods of Idiopathic Intracranial Hypertension
Brief Title: Current Treatment Methods of Idiopathic Intracranial Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Mansour, Doctor, Assiut University
Other Study IDs: treatment methods of IIH
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: IIH - Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lumbar puncture — Medical treatment Lumbar puncture Theco peritoneal shunt
  Other Names: Theco peritoneal shunt

SUMMARY:
Aim of the study :

1. to determine the response to each treatment plan.
2. to determine when to choose specific treatment method.
3. to determine complication of each type of treatment method

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) is caused by an elevation of intracranial pressure (ICP). The condition mainly affects obese young women of childbearing age.

In a recent study in the United Kingdom University of Kentucky urokinase, the estimated annual incidence was 4.7 % which represents a growth of 108% in 14 years, and parallels the growth of obesity prevalence .

The combination of raised intracranial pressure, without hydrocephalus or mass lesion, normal cerebrospinal fluid (CSF) composition and where no underlying aetiology is found are accepted criteria for the diagnosis of IIH.

The two most prominent symptoms of IIH are progressive visual deterioration and chronic headache, although additional symptoms including cranial nerve palsies, cognitive deficits, tinnitus and olfactory dysfunction are frequently also part of the clinical presentation. While the visual dysfunction is known to largely result from a pressure-induced papilledema, the origin of the IIH-related headache is less clear and therapeutic approaches are less investigated.

The conventional treatment for IIH involves weight loss, steroids, diuretics, and serial lumbar punctures and surgical treatment.

Surgical intervention should be conducted as soon as medical treatment fails. It is not acceptable to delay the intervention for patient with sever visual deterioration . Therefore surgery is indicated once visual loss continues despite optimum medical therapy .

Medical treatment with acetazolamide and serial lumbar punctures represent the initial management, in such cases preserving surgery to non-responding cases and those who cannot tolerate medical treatment.

Surgical treatment include lumboperitoneal shunt insertion , navigation guided ventriculo-peritoneal shunt ,endovascular stenting of sinuses in cases of sinus thrombosis and stenosis .

ELIGIBILITY:
Inclusion Criteria:

* patient has symptoms of increased intracranial pressure with :-

  * papilledema,
  * normal neurological examination,(except 6th nerve palsy),
  * elevated opening pressure( >=25 cm) csf,
  * normal csf content

Exclusion Criteria:

* Any patient diagnosed with increased intracranial pressure due to:

  * sinus thrombosis or stenosis will be excluded from this study and .accordingly endovascular stenting as a method of treatment will be excluded from this study.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients have symptoms of increased intracranial hypertension presenting to Assiut University hospital
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Patient improvement regarding headache, visual symptoms | 1 year
  Determine the Severity of headache on scale from (0-10) ((0-4)>mild, (5-7)>moderate, (8-10)>sever)
Patients improvement regarding fundus examination during regular visual assessment | 1 year
  Fundus examination grading (1-2-3-4)
Complication | 1 year
  Complication of each treatment option

SECONDARY OUTCOMES:
Other | 1 year
  Cost of treatment and hospital stay (Relation between type of treatment and cost Of treatment, time of hospital stay) (type of treatment and number of days of hospital stay)

CONTACTS AND LOCATIONS:
Overall Officials: Radwan Elnouby, Professor, Study Chair — Assiut University; Wael M Ali, AssProfessor, Study Director — Assiut University; Mohamed A Ragaee, AssProfessor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bubshait RF, Almomen AA. The Endonasal Endoscopic Management of Cerebrospinal Fluid Rhinorrhea. Cureus. 2021 Feb 20;13(2):e13457. doi: 10.7759/cureus.13457. PMID 33777546
- [Background] Mollan SP, Aguiar M, Evison F, Frew E, Sinclair AJ. The expanding burden of idiopathic intracranial hypertension. Eye (Lond). 2019 Mar;33(3):478-485. doi: 10.1038/s41433-018-0238-5. Epub 2018 Oct 24. PMID 30356129
- [Background] Friedman DI, Liu GT, Digre KB. Revised diagnostic criteria for the pseudotumor cerebri syndrome in adults and children. Neurology. 2013 Sep 24;81(13):1159-65. doi: 10.1212/WNL.0b013e3182a55f17. Epub 2013 Aug 21. PMID 23966248
- [Background] Markey KA, Mollan SP, Jensen RH, Sinclair AJ. Understanding idiopathic intracranial hypertension: mechanisms, management, and future directions. Lancet Neurol. 2016 Jan;15(1):78-91. doi: 10.1016/S1474-4422(15)00298-7. Epub 2015 Dec 8. PMID 26700907
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Akhter A, Schulz L, Inger HE, McGregor JM. Current Indications for Management Options in Pseudotumor Cerebri. Neurol Clin. 2022 May;40(2):391-404. doi: 10.1016/j.ncl.2021.11.011. Epub 2022 Mar 31. PMID 35465882